CLINICAL TRIAL: NCT02284243
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Evaluation of the Efficacy and Safety of Intranasal Dexmedetomidine for Postoperative Analgesia Following Bunionectomy
Brief Title: Placebo-Controlled Evaluation of Intranasal Dexmedetomidine for Postoperative Analgesia Following Bunionectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-14-013
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Pain, Post-operative
Keywords: Bunion; Bunionectomy; Pain; Analgesia; dexmedetomidine; intranasal
MeSH Terms: conditions — Pain, Postoperative; Bunion; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEX-IN 50mcg (Experimental): DEX-IN (Intranasal dexmedetomidine) 50mcg every 6 hours for 48 hours.
  Interventions: Drug: Intranasal Dexmedetomidine
- IN Placebo (Placebo Comparator): IN Placebo every 6 hours for 48 hours.
  Interventions: Drug: Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal Dexmedetomidine
  Other Names: DEX-IN
  Arms: DEX-IN 50mcg
Drug: Intranasal Placebo
  Arms: IN Placebo

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy, on Post-Operative Day (POD) 1, of DEX-IN compared with placebo, using the summed pain intensity difference over the first 48 hours (SPID48) in subjects with acute moderate to severe pain following unilateral bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent.
* Male or female between 18 and 70 years of age, inclusive.
* Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair
* Be American Society of Anesthesiology (ASA) physical class 1 or 2.
* Female subject are eligible only if all the following apply:

  * Not pregnant;
  * Not lactating;
  * Not planning to become pregnant during the study;
  * Be surgically sterile; or at least two year post menopausal; or have a monogamous partner who is surgically sterile; or is practicing double-barrier contraception; or practicing abstinence; or using an insertable, injectable, transdermal, or combination oral contraceptive.
* Male subjects must be surgically sterile or commit to the use of a reliable method of birth control
* Have a body mass index ≤35 kg/m2
* Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.

Exclusion Criteria:

* Have a known allergy to dexmedetomidine or any excipient in DEX-IN/placebo or to any peri- or postoperative medications used in this study.
* Have a clinically significant abnormal clinical laboratory test value.
* Have history of or positive test results for HIV, or hepatitis B or C.
* Have a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.
* Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.
* Have another painful physical condition that may confound the assessments of post operative pain.
* Have a history of syncope or other syncopal attacks.
* Have evidence of a clinically significant 12 lead ECG abnormality.
* Have a history of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) or prescription/illicit drug abuse..
* Have positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.
* Have a history or evidence of orthostatic hypotension.
* Have a resting heart rate of <50 beats per minutes or systolic blood pressure <100mmHg.
* Have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months.
* Use concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which in the investigator's opinion may exert significant analgesic properties or act synergistically with DEX-IN.
* Unable to discontinue medications, that have not been at a stable dose for at least 14 days prior to the scheduled bunionectomy procedure, within 5 half lives of the specific prior medication (or, if half life is not known, within 48 hours) before dosing.
* Have utilized any intranasal medications within the preceding 10 days.
* Have signs or a history of significant rhinitis or rhinorrhea (constant or chronic), nasal polyps, mucosal lesions of the nostril, postnasal drip of any etiology (constant or chronic), nasal ulcers, septal perforation or deviation, any nasal surgery, anosmia, nasal piercings, or frequent nosebleeds or other nasal pathology, that is sufficient to interfere with IN drug delivery.
* Have had an upper respiratory tract infection within 14 days of screening.
* Have utilized corticosteroids, either systemically, inhalational either intranasally or oral, or by intra-articular injection, within 14 days prior to the study.
* Have received any investigational product within 30 days before dosing with study medication.
* Have previously received DEX-IN in clinical trials, or had bunionectomy in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (3):
- United States (3):
  - Trovare Clinical Research, Inc., Bakersfield, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Endeavor Clinical Trials, P.A., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- DEX-IN 50mcg: DEX-IN (Intranasal dexmedetomidine) 50mcg every 6 hours for 48 hours.
  Intranasal Dexmedetomidine
- IN Placebo: IN Placebo every 6 hours for 48 hours.
  Intranasal Placebo
Period: Overall Study
Arm/Group | DEX-IN 50mcg | IN Placebo
Started | 84 | 84
Completed | 80 | 81
Not Completed | 4 | 3
Not completed — Lack of Efficacy | 3 | 3
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set - All subjects receiving at least one study dose
Groups:
- Total: Total of all reporting groups
Arm/Group | DEX-IN 50mcg | IN Placebo | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 81 | 163
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.37) | 44.0 (13.08) | 44.0 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 75 | 154
  Male | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 39 | 72
  Not Hispanic or Latino | 51 | 45 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 21 | 41
  White | 59 | 56 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 84 | 84 | 168
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (4.31) | 27.4 (4.08) | 27.0 (4.20)
Baseline pain intensity score (NPRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was recorded using a Numeric Rating Scale (Range 0-10) where 0 equates to no pain, and 10 equates to the worst pain imaginable.
  units on a scale | 6.4 (1.42) | 6.7 (1.90) | 6.5 (1.68)

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Difference Over the First 48 Hours (SPID48).
Description: Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 0.25, 0.5, 0.75, 1, 2, 4, and 6 hours post Dose 1. Thereafter pain assessments were to be recorded every 2 hours until 48 hours post Dose 1. Pain intensity differences from baseline were calculated at each time point and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation.
Time Frame: 48 hours
Population: mITT population, including all randomized subjects who received at least one study dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 84 | 84
units on a scale | -2328.2 (5746.724) | -548.90 (5819.373)
Statistical Analysis 1: Comparison: DEX-IN 50mcg vs IN Placebo; Test type: Superiority or Other; p = 0.0180, ANCOVA

2. Secondary Outcome: SPID at Various Other Time Points
Description: as for outcome 1
Time Frame: Up to 48 Hours
Population: mITT population, including all randomized subjects who received at least one study dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 84 | 84
units on a scale
  SPID 0-6 | -346.57 (579.0378) | -120.46 (590.7313)
  SPID 0-12 | -568.89 (1213.410) | -151.93 (1263.656)
  SPID 0-24 | -1043.2 (2553.890) | -239.07 (2717.394)
Statistical Analysis 1: Comparison: DEX-IN 50mcg vs IN Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA — Applies to SPID 0-6, SPID 0-12, and SPID 0-24

3. Secondary Outcome: Time to Perceptible and Meaningful Pain Relief
Description: Kaplan-Meier analysis of time to perceptible and meaningful pain relief for 50th percentile of subjects. Time to perceptible pain relief and time to meaningful pain relief were measured using the double-stopwatch method. The first stopwatch was given to each subject with the instructions to stop the watch when they first perceive pain relief to occur (time to perceptible relief). Once the first watch was stopped, the second stopwatch was given to the subject with the instructions to stop the watch when they are first experiencing meaningful pain relief (time to meaningful relief). A shorter time to pain relief is better.
Time Frame: 6 hours
Population: mITT population, including all randomized subjects who received at least one study dose
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 84 | 84
minutes
  Time to perceptible pain relief | 18.39 [15.50 to 25.68] | 33.0 [18.18 to 85.33]
  Time to meaningful pain relief | 79.32 [55.25 to 151.88] | NA [NA to NA] — Sufficient number of subjects did not achieve endpoint for analysis
Statistical Analysis 1: Comparison: DEX-IN 50mcg vs IN Placebo; Test type: Superiority or Other; p < 0.05, Log Rank — Applies to perceptible and meaningful pain relief

4. Secondary Outcome: Number of Subjects With Significant Pain Improvement Following the First Study Dose.
Time Frame: 6 hours
Population: mITT population, including all randomized subjects who received at least one study dose
Measure: Number; unit: participants
Arm/Group | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 84 | 84
participants
  ≥30% reduction in pain | 26 | 15
  ≥50% reduction in pain | 9 | 2
Statistical Analysis 1: Comparison: DEX-IN 50mcg vs IN Placebo; Test type: Superiority or Other; p < 0.05, Cochran-Mantel-Haenszel — Applies to ≥30% and ≥50% reduction in pain; Test for general association stratified by site

5. Secondary Outcome: Use of Rescue Medication (Oral Opioids)
Description: Number of subjects requiring rescue medication (Oral opioids) within 48 hours after first study dose
Time Frame: 48 hours
Population: mITT population, including all randomized subjects who received at least one study dose
Measure: Number; unit: participants
Arm/Group | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 84 | 84
participants | 66 | 76

6. Secondary Outcome: Time to First Rescue Medication Use
Description: Kaplan Meier analysis of time to first use of rescue analgesia 50th percentile of subjects. Rescue analgesia (oral oxycodone) was available to subjects with inadequately controlled pain. All doses of rescue analgesia administered were recorded and the time from the first study dose to first rescue analgesia in each subject was evaluated. A longer time to first rescue is better.
Time Frame: 48 hours
Population: mITT population, including all randomized subjects who received at least one study dose
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 84 | 84
hours | 4.94 [4.03 to 7.85] | 2.68 [1.42 to 3.47]
Statistical Analysis 1: Comparison: DEX-IN 50mcg vs IN Placebo; Test type: Superiority or Other; p = 0.0009, Log Rank

7. Secondary Outcome: Number of Subjects With Complete Protection From PONV
Time Frame: 24 hours
Population: mITT population, including all randomized subjects who received at least one study dose
Measure: Number; unit: participants
Arm/Group | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 84 | 84
participants | 72 | 70
Statistical Analysis 1: Comparison: DEX-IN 50mcg vs IN Placebo; Test type: Superiority or Other; p = 0.7718, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: All AEs were collected through the Day 7 study visit. All SAEs were assessed through the Day 7 visit, but were reported through 30 days of the last study visit if the investigator was made aware of the event.
Arm/Group | DEX-IN 50mcg | IN Placebo
Serious Adverse Events (participants affected / at risk) | 1/84 | 0/84
Other Adverse Events (participants affected / at risk) | 51/84 | 36/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEX-IN 50mcg (N=84) | IN Placebo (N=84)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEX-IN 50mcg (N=84) | IN Placebo (N=84)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (14) | 14 (15)
Vomiting (Gastrointestinal disorders) | 4 (5) | 6 (6)
Incision Site Erythema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood Pressure Decreased (Investigations) | 22 (22) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.